CLINICAL TRIAL: NCT03546829
Title: Safety Trial of Antimicrobial Therapy and Precision Radiation Therapy in Patients With Oligoprogressive Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 08517; 827551 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Early Stage Non-Small Cell Lung Cancer
MeSH Terms: interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 - Experimental (Experimental): Patients planned to undergo precision hypofractionated radiation to all sites of oligoprogression will receive vancomycin for 1 week before RT and for 1 month after start of RT, and asked to provide stool and blood samples as outlined in the Safety Trial study table.
  Interventions: Drug: Vancomycin; Radiation: Precision hypofractionated radiation

INTERVENTIONS:
Drug: Vancomycin — 125 mg, 4x daily for 5 weeks
Radiation: Precision hypofractionated radiation — Patients planned to undergo precision hypofractionated radiation to all sites of oligoprogression and will receive vancomycin for 1 week before RT and for 1 month after start of RT, and asked to provide stool and blood samples as outlined in the Safety Trial study table.

SUMMARY:
The first phase of this study was an open label, randomized pilot study. Enrollment for this phase is now complete.

The second phase is a single arm phase 1 safety study. Patients planned to undergo precision hypofractionated radiation to all sites of oligoprogression will receive vancomycin for 1 week before RT and for 1 month after start of RT, and asked to provide stool and blood samples as outlined in the Safety Trial study table.

ELIGIBILITY:
Randomized Pilot Inclusion

* Patients planned to receive Stereotactic Body Radiotherapy (SBRT) to a biopsy-proven or clinically-suspected NSCLC
* Age >18 years' old
* Patient capable of giving informed consent

Randomized Pilot Exclusion

* Use of antibiotics, antifungal, antivirals or antiparasitics during the 4 weeks prior to registration
* Active infection with oral temperature >100°F
* Use of corticosteroids, methotrexate or immunosuppressive drugs during the 4 weeks prior to registration
* Use of chemotherapy during the 4 weeks prior to radiotherapy or during radiotherapy. Chemotherapy cannot begin before the collection of the 30-day post treatment sample (S4).
* Documented history of HIV, HBV or HCV
* Active uncontrolled gastrointestinal disorders such as inflammatory bowel disease, moderate/severe irritable bowel syndrome, persistent, infectious gastroenteritis, colitis or gastritis, persistent or chronic diarrhea of unknown etiology, Clostridium Difficile infection (within 2 years of lung cancer diagnosis) or Helicobacter Pylori infection (untreated)
* Major surgery of the GI tract, with the exception of cholecystectomy and appendectomy, in the past five years. Any major bowel resection at any time
* Patients on anti-diarrheal medications
* Patients on probiotics

Safety Trial Inclusion

* Patients planned to receive precision hypofractionated radiation (SBRT or an ablative dose of radiation is used if SBRT is not appropriate or if insurance does not approve - i.e. > 30 Gy in 10 fraction equivalent) to all sites of oligoprogressive NSCLC who progressed after 1st line systemic therapy for metastatic disease which included immunotherapy or a tyrosine kinase inhibitors (TKI) for NSCLC
* The number of sites of progression are < 5 sites.
* Age >18 years' old
* Patient capable of giving informed consent

Safety Trial Exclusion

* Evidence of untreated CNS or leptomeningeal disease
* Use of antibiotics, antifungal, antivirals or antiparasitics during the 4 weeks prior to registration
* Active infection with oral temperature >100°F
* Use of oral corticosteroids, methotrexate or immunosuppressive drugs during the 4 weeks prior to registration
* Use of chemotherapy during the 4 weeks prior to radiotherapy or during radiotherapy. Chemotherapy cannot begin before the collection of the 30-day post treatment sample (S3).
* Documented history of HIV, HBV or HCV
* Patients on daily anti-diarrheal medications
* Use of probiotics during the 4 weeks prior to radiotherapy or during radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-03-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Randomized Pilot: Th1 immune response measured by cytokine expression (IFN gamma). | 2 years
  The primary endpoint is IFN-gamma cytokine expression at Day 30 (+/- 2) collection compared to the pre-radiation level. It will be analyzed using generalized linear mixed models.
Randomized Pilot: the safety of the addition of vancomycin to Stereotactic Body Radiotherapy | 2 years
  The primary safety endpoint is uncontrolled diarrhea, as defined by CTCAE v4.0 > or = grade 3 (Increase of >=7 stools per day over baseline; incontinence; hospitalization indicated; severe increase in ostomy output compared to baseline; limiting self-care ADL). This will be evaluated during treatment and at 1 month, 3 months, 6 months and 12 months.
Safety Trial: the safety of the addition of vancomycin to precision hypofractionated radiation | 3 years
  Safety Trial: The primary safety endpoint is uncontrolled diarrhea, as defined by CTCAE v5.0 > or = grade 3 Increase of >=7 stools per day over baseline; hospitalization indicated; severe increase in ostomy output compared to baseline; limiting self care ADL). This will be evaluated weekly during vancomycin use and RT, at 1 month post-vancomycin, 3 months post-vancomycin, 6 months post-vancomycin and 12 months post-vancomycin.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Feigenberg, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Feigenberg SJ, Costabile F, Tanes C, Bittinger K, O'Connor R, Agarwal D, Skoufos G, Salaris S, Hatzigeorgiou A, Kostopoulos N, Lloyd S, Friedes C, Chen L, Yegya-Raman N, Cengel K, Levin W, Valentic B, Quarton T, Shestov AA, Berman A, Bradley J, Maity A, Koumenis C, Ben-Josef E, Facciabene A. Enhancing outcomes in medically inoperable early-stage NSCLC with gut-targeted antibiotics and stereotactic body radiotherapy: results from a randomized pilot study. J Immunother Cancer. 2025 Jul 10;13(7):e011356. doi: 10.1136/jitc-2024-011356. PMID 40639850